CLINICAL TRIAL: NCT06838481
Title: Effects of Overload Eccentric and Concentric Resistance Training on the Cost of Walking, Muscle-tendon and Jumping Performance in Healthy Older Individuals
Acronym: EOECORT-COM-JP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hungarian University of Sports Science (Other)
Collaborators: Semmelweis University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelaziz Emam, PhD Student Semmelweis University, Hungarian University of Sports Science
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TE-KEB/No11/2024; TE-KEB/No11/2024 (Other: Hungarian University of sports science)
Record Dates: First submitted 2025-02-09; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Healthy Older Adults
Keywords: Resistance training; cost of walking; cost of transfer; balance; countermovement jump; SSC

STUDY DESIGN:
Intervention Model Description: Cross-Sectional Component:
  Purpose: To assess baseline muscle-tendon function, metabolic function, and other relevant measures in older adults.
  Design: Observational, providing a snapshot of the participants' characteristics before the intervention.
  Longitudinal Intervention Component:
  Purpose: To examine the effects of different training interventions over time and assess retention effects.
  Design: A three-arm parallel-group randomized controlled trial (RCT) with pre- and post-intervention assessments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Concentric overload resistance training (Active Comparator): Receive Concentric overload resistance training
  Interventions: Other: Concentric overload resistance training
- Eccentric overload resistance training (Experimental): Receive Eccentric overload resistance training
  Interventions: Other: Eccentric overload resistance training
- Active control group (Placebo Comparator): walking intervention
  Interventions: Other: Active Control

INTERVENTIONS:
Other: Concentric overload resistance training — * Resistance training groups will train 2-3 times per week for 3 months using specialized TechnoGym machines.
  * Exercises include Concentric leg press, knee extension, and ankle plantarflexion in a progressive loading program following American College of Sports Medicine (ACSM) & National Strength and Conditioning Association (NSCA) guidelines.
  * Heart rate, blood pressure, and perceived exertion will be monitored during each session.
  Other Names: active control
  Arms: Concentric overload resistance training
Other: Eccentric overload resistance training — * Resistance training groups will train 2-3 times per week for 3 months using specialized TechnoGym machines.
  * Exercises include Eccentric leg press, knee extension, and ankle plantarflexion in a progressive loading program following American College of Sports Medicine (ACSM) & National Strength and Conditioning Association (NSCA) guidelines.
  * Heart rate, blood pressure, and perceived exertion will be monitored during each session.
  Arms: Eccentric overload resistance training
Other: Active Control — Walking
  Arms: Active control group

SUMMARY:
Normal aging leads to a decline in neuromuscular and mobility functions, including a 60% reduction in maximal voluntary force production, a 25% decrease in muscle volume and quality (sarcopenia), and reduced tendon stiffness by age 70. These changes impair walking speed, balance, and increase the metabolic cost of walking by ~20% in older adults compared to younger individuals. While walking training can reduce metabolic costs, no interventions have successfully addressed the 20% age-related difference. Resistance training, particularly eccentric (muscle-lengthening) training, shows promise for improving muscle strength and mass, but its effects on functional, cognitive abilities, and walking economy in older adults remain unexplored.

DETAILED DESCRIPTION:
Normal aging is characterized by a decline in neuromuscular and mobility functions. By the age of 70, maximal voluntary force production decreases by approximately 60%, accompanied by a ~25% reduction in muscle volume and quality, leading to sarcopenia. Alongside changes in muscle protein content, composition, and mitochondrial biochemistry, aging also affects tendon properties. While healthy aging does not significantly alter tendon size, it reduces tendon stiffness, which can delay force transmission. These changes in muscle-tendon function contribute to slower walking speeds and impaired static and dynamic balance.

One of the most significant functional changes with aging is the increased metabolic cost of walking. Older individuals require ~20% more metabolic energy to walk the same distance as younger adults, yet the underlying reasons remain unclear. While walking training has been shown to reduce metabolic costs in older adults, no studies have attempted to reduce this 20% age-related difference using alternative interventions.

Resistance training induces adaptations in muscle-tendon function by requiring participants to overcome external loads. Traditional resistance training combines concentric (muscle shortening) and eccentric (muscle lengthening) contractions, but eccentric training has received increasing attention due to its superior benefits in muscle strength and mass improvement. However, no studies have examined how resistance training, particularly with an eccentric focus, impacts functional and cognitive abilities or walking economy in older adults.

Objectives:

This study aims to:

1. Investigate the effects of resistance training, particularly eccentric-focused training, on muscle-tendon function and walking economy in older adults.
2. Examine whether these changes translate into improved neuromuscular and cognitive functions.
3. Determine if improved tendon stiffness leads to more efficient force transmission, reducing walking energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy men and women aged 60+ (intervention study).

  * No significant cognitive or cardiovascular impairments.

Exclusion Criteria:

* • Acute injuries or history of severe tendon injuries (Achilles or patellar tendon rupture).

  * Tendinopathy or chronic musculoskeletal disorders.
  * Hypertension, unless controlled with medication.
  * Neurological or psychiatric disorders (dementia, mild cognitive impairment).
  * Metabolic diseases affecting muscle/tendon function,

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Walking metabolic cost | Through study completion, an average of 1.5 year
  Assessed using spirometry at different speeds (J/kg/m)

SECONDARY OUTCOMES:
Maximum isometric voluntary contraction | Through study completion, an average of 1.5 year
  Maximum isometric voluntary force using a dynamometer. (Nm)
Patella and Achilles tendon stiffness | Through study completion, an average of 1.5 year
  Stiffness is the slope of the force elongation curve using dynamometer combining with Ultrasound (N/mm)
Vastus lateralis and Gastrocnemius muscle thickness & tendon thickness | Through study completion, an average of 1.5 year
  VL, GC, and Achilles tendon & patellar tendon will be assessed using Ultrasound images (mm)
Whole leg muscle mass | Through study completion, an average of 1.5 year
  Whole leg muscle mass via DEXA scan.(Kg)
Jump efficiency | Through study completion, an average of 1.5 year
  squat jump and Countermovement jump height (cm) jump efficiency (%)
Cognitive Assessments | Through study completion, an average of 1.5 year
  Cognitive tests: Executive function, working memory, and processing speed using some questionnaires with score values.
  Reaction Time (milliseconds, ms) Score (points or errors) - Based on correct/incorrect responses in tasks Number of correct responses per second (responses/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. DR. Tibor Hortobágyi Hortobágyi, Principal Investigator — Hungarian University of Sports Science, Department of Kinesioogy, Budapest, Hungary
Locations (1):
- Hungarian University of Sports Science, Budapest, Hungary, Budapest XII., Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 15 May 2026

REFERENCES:
- [Background] Malatesta D, Canepa M, Menendez Fernandez A. The effect of treadmill and overground walking on preferred walking speed and gait kinematics in healthy, physically active older adults. Eur J Appl Physiol. 2017 Sep;117(9):1833-1843. doi: 10.1007/s00421-017-3672-3. Epub 2017 Jul 7. PMID 28687953
- [Background] Thomas EE, De Vito G, Macaluso A. Speed training with body weight unloading improves walking energy cost and maximal speed in 75- to 85-year-old healthy women. J Appl Physiol (1985). 2007 Nov;103(5):1598-603. doi: 10.1152/japplphysiol.00399.2007. Epub 2007 Sep 6. PMID 17823302
- [Background] Valenti G, Bonomi AG, Westerterp KR. Multicomponent Fitness Training Improves Walking Economy in Older Adults. Med Sci Sports Exerc. 2016 Jul;48(7):1365-70. doi: 10.1249/MSS.0000000000000893. PMID 26848888
- [Background] Hunter GR, Fisher G, Neumeier WH, Carter SJ, Plaisance EP. Exercise Training and Energy Expenditure following Weight Loss. Med Sci Sports Exerc. 2015 Sep;47(9):1950-7. doi: 10.1249/MSS.0000000000000622. PMID 25606816
- [Background] Hunter GR, McCarthy JP, Bryan DR, Zuckerman PA, Bamman MM, Byrne NM. Increased strength and decreased flexibility are related to reduced oxygen cost of walking. Eur J Appl Physiol. 2008 Nov;104(5):895-901. doi: 10.1007/s00421-008-0846-z. Epub 2008 Aug 29. PMID 18758805
- [Background] Godges JJ, MacRae PG, Engelke KA. Effects of exercise on hip range of motion, trunk muscle performance, and gait economy. Phys Ther. 1993 Jul;73(7):468-77. doi: 10.1093/ptj/73.7.468. PMID 8316580